CLINICAL TRIAL: NCT03446963
Title: Feasibility Study of the Groups for Health Intervention for Adults Accessing Treatment for Depression
Brief Title: Social Connectedness Group Intervention in Depression
Acronym: G4H-A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 17110
Record Dates: First submitted 2018-02-14; First posted 2018-02-27 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Population Groups; Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm: Groups 4 Health (Experimental): Social group intervention. The aim is to practice participating in a social group within a safe environment; to identify groups and social networks which are meaningful for the person; and to understand any barriers people may have to engaging with these groups/networks.
  Interventions: Behavioral: Groups for Health

INTERVENTIONS:
Behavioral: Groups for Health — Group sessions, 5 modules x 1.5 hours (once per week). Modules focus on psychoeducation, mapping existing social networks, examining barriers to engagement in existing networks, goal setting and identifying new groups to join.

SUMMARY:
This study evaluates the feasibility of the Groups for Health (G4H) intervention for adults accessing support for depression in the UK. G4H targets improvements in adults' interpersonal functioning in order to reduce feelings of loneliness. The study will adapt the G4H intervention for delivery to adults seeking treatment for depression in the UK and estimate trial parameters (recruitment, retention, missing data and acceptability) of the adapted intervention, prior to a definitive trial. A mixed methods design of interviews and a single group, pre-post study will be employed.

DETAILED DESCRIPTION:
Background: Loneliness is frequently reported amongst adults with depression. Interventions to reduce loneliness in different populations have shown mixed results. The Groups for Health (G4H) programme has been developed according to the social identity approach within social psychology and has demonstrated preliminary efficacy for reducing loneliness in a proof-of-concept study conducted with Australian student sample. The present study will examine whether G4H can be adapted to suit the needs of a clinical population in the context of UK secondary care services.

Objective: Phase 1 - To adapt the G4H intervention for delivery to adults seeking treatment for depression in the UK. Phase 2: To estimate trial parameters (recruitment, retention, missing data and acceptability) of the adapted intervention, prior to a definitive trial; to optimise the adapted intervention for delivery to adults accessing treatment for depression in the UK; to optimise evaluation procedures (candidate outcome measures)

Trial configuration: sequential exploratory mixed methods design. Phase 1: one-to-one interviews. Phase 2: Activity 1 (intervention), single group, pre-post study. Activity 2 (interviews): one-to-one interviews.

Condition: Depression

Interventions: group-based behavioural programme

ELIGIBILITY:
Inclusion Criteria:

Phase 1

Service user participants:

* Aged 18-65
* Accessing treatment for depression
* Loneliness: score 6 or above on the University of California Loneliness Scale (UCLA-3) (Hughes et al., 2004)
* Able to speak/read English
* Ability to give informed consent

Staff participants:

- Clinical practitioner with at least 6 months experience of working with people with depression

Phase 2 Activity 1: intervention

* Aged 18-65
* Accessing treatment for depression
* Loneliness: score 6 or above on the University of California Loneliness Scale (UCLA-3) (Hughes et al., 2004)
* Able to speak/read English
* Ability to give informed consent

Activity 2: interviews

- Attended or agreed to attend Phase 2, Activity 1

Exclusion Criteria:

* None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-03-18 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment | 3 months
  The proportion of patients contacted for screening against those who are consented
Feasibility of enrollment | 3 months
  The proportion of patients consented against those enrolled
Feasibility of data collection | 8 weeks
  The overall proportion of survey measures completed by each participant at each of the 2 time points
Patient retention | 8 weeks
  The proportion of patients attending all five G4H sessions

CONTACTS AND LOCATIONS:
Overall Officials: Tom Dening, MD, Study Chair — University of Nottingham
Locations (1):
- Nottinghamshire Healthcare NHS Foundation Trust, Nottingham, Nottinghamshire, United Kingdom

REFERENCES:
- [Background] Baker SL, Heinrichs N, Kim HJ, Hofmann SG. The liebowitz social anxiety scale as a self-report instrument: a preliminary psychometric analysis. Behav Res Ther. 2002 Jun;40(6):701-15. doi: 10.1016/s0005-7967(01)00060-2. PMID 12051488
- [Background] Hays RD, DiMatteo MR. A short-form measure of loneliness. J Pers Assess. 1987 Spring;51(1):69-81. doi: 10.1207/s15327752jpa5101_6. PMID 3572711
- [Background] Hughes ME, Waite LJ, Hawkley LC, Cacioppo JT. A Short Scale for Measuring Loneliness in Large Surveys: Results From Two Population-Based Studies. Res Aging. 2004;26(6):655-672. doi: 10.1177/0164027504268574. PMID 18504506
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Van Orden KA, Cukrowicz KC, Witte TK, Joiner TE. Thwarted belongingness and perceived burdensomeness: construct validity and psychometric properties of the Interpersonal Needs Questionnaire. Psychol Assess. 2012 Mar;24(1):197-215. doi: 10.1037/a0025358. Epub 2011 Sep 19. PMID 21928908